CLINICAL TRIAL: NCT05829967
Title: Chemotherapy Induced Peripheral Neuropathy (CIPN ) and it's Impact on Quality of Life in Patients Receiving Platinum and Taxanes at Assuit University Hospital
Brief Title: CIPN and it's Impact on Quality of Life in Patients Receiving Platinum and Taxanes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Khalifa Fathy, Principal Investigator, Assiut University
Other Study IDs: CIPN
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Neuropathies are a major cause of moderate to severe impairments in cancer patients.

Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most frequent side effects caused by antineoplastic agents, with a prevalence from 19% to over 85%.

DETAILED DESCRIPTION:
Neuropathies are a major cause of moderate to severe impairments in cancer patients .

Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most frequent side effects caused by antineoplastic agents, with a prevalence from 19% to over 85%.

There are six main substance groups that cause damage to neurons developing CIPN: platinum-based antineoplastic agents, vinca alkaloids, epothilones (ixabepilone), taxanes, proteasome inhibitors (bortezomib) and immunomodulatory drugs (thalidomide).

Platinum-based chemotherapeutics (oxaliplatin, cisplatin and carboplatin) have the highest prevalence rates of CIPN, affecting ~ 70% of patients, often complicated by coasting Acute oxaliplatin-induced peripheral neuropathy (OIPN) can result in prolonged infusion times (~ 22%), dose reduction (15-43%) and treatment cessation (6-21.4%) Taxane-induced peripheral neuropathy (TIPN) (paclitaxel, Docitaxel and Cabazitaxel ) is the most common non-haematological adverse event of treatment,however, docetaxel is generally considered to be less neurotoxic than paclitaxel.

CIPN occurs in a dose-dependent manner usually ,duration of exposure, scheduling and combination therapies are also potential risk factors.

diabetes mellitus and increasing age (≥75 years) have been proposed as strong independent risk factors(9). In addition to ,alcohol abuse, renal insufficiency, hypothyroidism, infections like (HIV) and smoking.

The severity of neuropathies can be graded by (Grading scales of CIPN includes; National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Most commonly used , WHO grading system ,self-assessment by patients is preferable due to consistent underrating by healtcare professionals.

symptoms of CIPN in hands and feet, such as tingling, numbness, cramps can cause problems with regular daily activities , standing and walking , Patients became limited in their daily activities and number of them stated that they became more dependent on others.

Treatment strategies depends on discontinuation or lowering the dose . Persistent neuropathic pain can be treated with anti-seizure medications, antidepressants, or analgesics . In severe painful conditions patients may be referred to the Chronic Pain Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and <75 .
* Sex : Male or female
* Adjuvant or metastatic
* Receiving neurotoxic agents " platinum and taxanes "
* No documentation of any other causes of neuropathy in their medical records as : congenital and DM

Exclusion Criteria:

* Pt not receiving any neurotoxic CTH.
* Detected other causes of neuropathy.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 cases aged 18 years to 75 years who receiving taxanes and platinum
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with CIPN who receiving taxanes and platinum | Baseline
  Number of patients with CIPN who receiving taxanes and platinum compounds in different chemotherapy regimens
Rae of recovery in patients with CIPN who receiving taxanes and platinum | Baseline
  Possibility of recovery in patients with CIPN who receiving taxanes and platinum compounds in different chemotherapy regimens and assessment by nerve conduction test.

CONTACTS AND LOCATIONS:
Overall Officials: Taha Zaki, Prof, Principal Investigator — Assiut University; Mohamed Alaa El Deen, Assist prof, Principal Investigator — Assiut University; Samar El Morshidy, Assist prof, Principal Investigator — Assiut University